CLINICAL TRIAL: NCT06095518
Title: DIC Markers and Thrombin Generation Parameters in Patients on ECMO Support: a Pilot Study
Acronym: DIC-ECMO
Status: Recruiting | Type: Observational
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Wincy Wing-Sze Ng, Associate Consultant, Adult Intensive Care Unit, Queen Mary Hospital, Hong Kong
Other Study IDs: UW 23-259
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-10

CONDITIONS: Extracorporeal Circulation; Complications; Extracorporeal Membrane Oxygenation Complication
Keywords: ECMO; Thrombosis; Haemorrhage
MeSH Terms: conditions — Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Adult Intensive Care Unit, Queen Mary Hospital
  Interventions: Diagnostic Test: DIC markers and Thrombin Generation Parameters
- Department of Intensive Care Unit, Tuen Mun Hospital
  Interventions: Diagnostic Test: DIC markers and Thrombin Generation Parameters

INTERVENTIONS:
Diagnostic Test: DIC markers and Thrombin Generation Parameters — Observation of DIC markers and thrombin generation parameters in patients with and without thrombotic and hemorrhagic complications

SUMMARY:
To study the correlation between novel DIC markers and thrombin generation parameters with thrombotic and hemorrhagic complications of patients on ECMO support.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18; AND
* Admitted to the mixed medical-surgical intensive care units of Queen Mary Hospital or Tuen Mun Hospital in Hong Kong; AND
* Require either veno-arterial (VA) or veno-venous (VV) extracorporeal membrane oxygenation (ECMO) support.

Exclusion Criteria:

* Patients who are on central VA-ECMO support; OR
* Patients with missing clinical data; OR
* Patients with pre-existing thromboembolism requiring long term anticoagulation prior to ECMO cannulation; OR
* Post-operative admissions

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring ECMO support
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of thrombotic and hemorrhagic events | From the start of ECMO support to the end of ECMO support (which can be variable, typically around 5 days to 1 week)
  Thrombotic events include circuit-related thrombosis (e.g. oxygenator failure requiring circuit change) OR Non-circuit-related thrombosis (e.g. new pulmonary embolism or deep vein thrombosis while on ECMO.
  Hemorrhagic events include bleeding at critical sites or requiring interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided